CLINICAL TRIAL: NCT00107796
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of PROVIGIL ® (Modafinil) Treatment (100, 200, and 400 mg/Day) in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy
Brief Title: Study of PROVIGIL ® (Modafinil) Treatment in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1538/3027/NA/MN-Narcolepsy
Record Dates: First submitted 2005-04-08; First posted 2005-04-11 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2006-05

CONDITIONS: Narcolepsy
Keywords: Pediatric Narcolepsy; Excessive sleepiness
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
Primary Objectives: The primary objectives of the study are to determine the effectiveness of PROVIGIL treatment, compared to placebo treatment, in children and adolescents with excessive sleepiness (ES) associated with narcolepsy, as assessed by:

* mean sleep latency from the Multiple Sleep Latency Test (MSLT) (average of 4 naps performed at 0900, 1100, 1300, and 1500) at the last post-baseline observation (week 6 or early termination)
* the Clinical Global Impression of Change (CGI-C) ratings for ES, at the last post-baseline observation (week 6 or early termination).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis and Main Criteria for Inclusion (Patients are included in the study if all of the following criteria are met):

* Written informed consent/assent is obtained
* A boy or girl aged 6 through 16 years, inclusive
* Meet the minimal criteria established by the International Classification of Sleep Disorders (ICSD) manual of the American Academy of Sleep Medicine (AASM) for narcolepsy (or presumed narcolepsy) as assessed by all of the following: *clinical history;

  * NPSG (nocturnal polysomnogram) (as evaluated by the investigator) to rule out other sleep disorders (ie, obstructive sleep apnea/hypopnea syndrome [OSAHS] or periodic limb movement with sleep [PLMs]);
  * narcolepsy (or presumed narcolepsy) as identified by at least 1 of the following: MSLT (as evaluated by the investigator) (mean sleep latency [from 4 naps] <10 minutes); 2 sleep onset REM periods (SOREMP); cataplexy; sleep paralysis; hypnogogic hallucinations -OR- *have a previous diagnosis of narcolepsy on the basis of NPSG and/or MSLT at any time before the screening visit
* Have ES (MSLT <10 minutes and/or CGI S ≥4) that is not a direct result of inadequate sleep hygiene or other medical disorder
* Are in good health as determined by a medical and psychiatric history, physical examination, ECG, and clinical laboratory tests
* Have blood pressure values greater than those for the 5th percentile and less than the 95th percentile for age on the National High Blood Pressure Education Program guidelines for blood pressure levels for boys and girls ages 6 through 16 years
* Girls who are post menarche or sexually active must have a negative urine pregnancy test prior to the baseline visit, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence.
* Be able to swallow a placebo tablet the same size and shape as the study drug tablet
* Negative UDS (urine drug screen) for any illicit drug, alcohol (ethanol), stimulants, or modafinil at screening; if positive for stimulants or modafinil (prescribed for ES) at the screening visit, UDS to be repeated after a washout period and before the baseline visit
* Have a parent or legal guardian who is willing to participate in the study

Exclusion Criteria:

Main Criteria for Exclusion (Patients are excluded from participating in this study if 1 or more of the following criteria are met):

* Have any other disorder(s) that could be considered the primary cause of ES (eg, self induced sleep deprivation)
* Have a past or present seizure disorder (except history of a single febrile seizure), a history of psychosis, or of clinically significant head trauma (eg, brain damage) or past neurosurgery
* Have a history of suicide attempt, or are at suicidal risk
* Have an average of 5 or more apneic/hypopneic episodes per hour of nocturnal sleep as assessed by NPSG at the baseline visit
* A clinically significant drug sensitivity to stimulants such as amphetamine, dextroamphetamine, methylphenidate, or pemoline; and/or modafinil or any of its components
* Use of any prescription (eg, clonidine, guanfacine) or nonprescription (over the counter [OTC]) medications, including dietary supplements with psychoactive properties (eg, any OTC medications or supplements containing ephedrine [ie, ma huang or ephedra], pseudoephedrine, caffeine, or phenylpropanolamine) or sedating properties (ie, antihistamines or sedative hypnotics) within 1 week of the baseline visit (Note: Medications for the treatment of cataplexy will be permitted if the patient has been on a stable dose for at least 1 month.)
* Use of any MAO (monoamine oxidase) inhibitors or SSRIs (Selective Serotonin Reuptake Inhibitors) within 2 weeks of the baseline visit (unless used for cataplexy)
* Received any investigational drug (except modafinil) within 4 weeks of the baseline visit
* Any disorder that could interfere with drug absorption, distribution, metabolism, or excretion (including previous gastrointestinal surgery)
* Active, clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other major clinically significant disorder/disease
* Any clinically significant deviation from the normal range(s) in the physical examination or ECG findings, or clinical laboratory test results (ie, serum chemistry, hematology, and urinalysis) at the screening or baseline visit
* ANC (absolute neutrophil count) below the lower limit of normal at the screening visit (Note: If the ANC is below the lower limit of normal at the baseline visit, the medical monitor will be consulted for continued eligibility in the study.)
* Seated pulse outside the range of 60 through 115 bpm after resting for 5 minutes
* A history of alcohol, narcotic, or any other substance abuse or dependence as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM IV) criteria
* A total daily intake of more than 250 mg of caffeine per day (eg, approximately five 12 ounce caffeinated sodas, 2.5 cups of coffee or tea, or about 12.5 ounces of chocolate per day) within 1 week of the baseline visit
* Pregnant or lactating/nursing girl; any girl who becomes pregnant during the study will be withdrawn
* A clinically significant illness within 4 weeks of the baseline visit; or is symptomatic for any clinically significant illness at the screening or baseline visit

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
Mean sleep latency from the Multiple Sleep Latency Test (MSLT) (average of 4 naps performed at 0900, 1100, 1300, and 1500) at the last post baseline observation (week 6 or early termination)
The Clinical Global Impression of Change (CGI-C) ratings for ES, at the last post baseline observation (week 6 or early termination)

SECONDARY OUTCOMES:
Clinical Global Impression of Change (CGI-C) ratings for ES at weeks 3 and 6
Total score from the Pediatric Daytime Sleepiness Scale (PDSS) at weeks 3 and 6, and last postbaseline observation
Mean sleep latency from the MSLT (average of 4 naps performed at 0900, 1100, 1300, and 1500) at week 6

CONTACTS AND LOCATIONS:
Locations (73):
- United States (68):
  - Robert Doekel, Jr., M.D., Birmingham, Alabama
  - Chris M. Makris, M.D., Birmingham, Alabama
  - Barbara Harris, Ph.D., Phoenix, Arizona
  - Derek Loewy, Ph.D., Tucson, Arizona
  - Stuart Quan, M.D., Tucson, Arizona
  - Joseph McCarty, M.D., Fort Smith, Arkansas
  - John L. Carroll, M.D., Little Rock, Arkansas
  - Samuel Boellner, M.D., Little Rock, Arkansas
  - Julie Thompson-Dobkin, D.O., Huntington Beach, California
  - Mark Buchfuhrer, M.D., Long Beach, California
  - Yury Furman, M.D., Los Angeles, California
  - Stuart Menn, M.D., Palm Springs, California
  - Richard Shubin, M.D., Pasadena, California
  - Lawrence Sher, M.D., Rolling Hills Estates, California
  - Milton K. Erman, M.D., San Diego, California
  - Stephen Brooks, M.D., San Francisco, California
  - Paul Haberman, M.D., Santa Monica, California
  - Jed Black, M.D., Stanford, California
  - Amerigo Padilla, M.D., Miami, Florida
  - Martin A. Cohn, M.D., Naples, Florida
  - D. Alan Lankford, Ph.D., Atlanta, Georgia
  - Gary Montgomery, M.D., Atlanta, Georgia
  - Jerry Silverboard, M.D., Atlanta, Georgia
  - Charles Wells, Jr., M.D., Macon, Georgia
  - Stephen H. Sheldon, D.O., FAAP, Chicago, Illinois
  - Michael Kohrman, M.D., Chicago, Illinois
  - Anna Ivanenko, M.D., Ph.D., Maywood, Illinois
  - Henry Lahmeyer, M.D., Northfield, Illinois
  - James Cook, M.D., Danville, Indiana
  - William Leeds, D.O., Topeka, Kansas
  - Karen Waters, M.D., Louisville, Kentucky
  - Margaret Ann Springer, M.D., Shreveport, Louisiana
  - Helene A. Emsellem, M.D., Chevy Chase, Maryland
  - Marc Raphaelson, M.D., Frederick, Maryland
  - Daniela Minecan, M.D., Ann Arbor, Michigan
  - George Zureikat, M.D., Flint, Michigan
  - John Harsh, Ph.D., DABSM, Hattiesburg, Mississippi
  - Pradeep Sahota, M.D., Columbia, Missouri
  - William Torch, M.D., MS, Reno, Nevada
  - Kathleen Ryan, M.D., Mount Laurel, New Jersey
  - Sushmita Mikkilineni, M.D., New Brunswick, New Jersey
  - Monroe Karetzky, M.D., Newark, New Jersey
  - Lee Brooks, M.D., Princeton, New Jersey
  - Marc Seelagy, M.D., Trenton, New Jersey
  - Gary Zammit, M.D., New York, New York
  - James Lee, M.D., Charlotte, North Carolina
  - Bruce Corser, M.D., Cincinnati, Ohio
  - Raouf Amin, MD, Cincinnati, Ohio
  - Martin Scharf, Ph.D., Cincinnati, Ohio
  - Carol Rosen, M.D., Cleveland, Ohio
  - Markus H. Schmidt, M.D., Ph.D., Dublin, Ohio
  - Michael Neeb, Ph.D., Toledo, Ohio
  - William C. Orr, Ph.D., Oklahoma City, Oklahoma
  - Jorg Pahl, M.D., Oklahoma City, Oklahoma
  - Dainis Irbe, M.D., Eugene, Oregon
  - William Pistone, M.D., Allentown, Pennsylvania
  - Jeffery Gould, M.D., Bethlehem, Pennsylvania
  - Guillermo Borrero, M.D., Clairton, Pennsylvania
  - Lee Brooks, M.D., Philadelphia, Pennsylvania
  - Judith Owens, M.D., MPH, Providence, Rhode Island
  - Richard Bogan, M.D., FCCP, Columbia, South Carolina
  - Julie Jacques, D.O., Morristown, Tennessee
  - John Hudson, M.D., Austin, Texas
  - David Sperry, M.D., Dallas, Texas
  - Todd J. Swick, M.D., Houston, Texas
  - Jerry J. Tomasovic, M.D., San Antonio, Texas
  - James M. Ferguson, M.D., Salt Lake City, Utah
  - Ralph A. Pascualy, M.D., Seattle, Washington
- Canada (5):
  - Adam Moscovitch, M.D., Calgary, Alberta
  - Leonid Kayumov, M.D., Scarborough Village, Ontario
  - Mortimer Mamelak, M.D., Toronto, Ontario
  - Colin Shapiro, Ph.D., Toronto, Ontario
  - Allen Denys, M.D., Windsor, Ontario

REFERENCES:
- See also: Related Info — http://www.sleeptrial.com